CLINICAL TRIAL: NCT04777461
Title: Living With Polycystic Ovary Syndrome- Structured Education Programme
Brief Title: Living With Polycystic Ovary Syndrome
Acronym: LW-PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: British Dietetic Association (Unknown)
Responsible Party: Principal Investigator, Thozhukat Sathyapalan, Professor/ Honorary consultant Endocrinologist, University of Hull
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LW-PCOS V1.2020
Record Dates: First submitted 2020-09-26; First posted 2021-03-02 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Pilot the structured education in women with PCOS
  Interventions: Other: Survey on patient's perspectives on the development of an structured education programme for PCOS; Other: Pre-pilot questionnaire; Other: Piloting the structured education programme for PCOS; Other: Post-pilot questionnaire; Other: cognitive outcomes outcome evaluation form

INTERVENTIONS:
Other: Survey on patient's perspectives on the development of an structured education programme for PCOS — The outcome of this survey will help with developing curriculum for the structured education programme.
Other: Pre-pilot questionnaire — The questionnaire is aimed to capture the knowledge and expectations of the participants from taking part in the educational sessions.
Other: Piloting the structured education programme for PCOS — Piloting the education program through 2 educational group sessions
Other: Post-pilot questionnaire — The questionnaire aimed to capture participant's satisfactions and knowledge gained by taking part in the pilot study
Other: cognitive outcomes outcome evaluation form — This aimed to capture skills developed, knowledge gained and changes in participants behaviour and perceptions by taking part in the pilot study.

SUMMARY:
This project aims to develop and pilot an evidence-based structured education program that can be run in groups to enable women with PCOS to make lifestyle changes, which will help them improve their PCOS and reduce the risk of future PCOS-related complications.

DETAILED DESCRIPTION:
The first aim of this project is to develop an evidence-based structured education programme for women with PCOS. According to the Medical Research Council framework for complex interventions, robust patient-education programmes should have an evidence-based structured written curriculum, which is delivered by trained educators and is regularly assessed and audited. To meet these standards, the investigators first aim to develop a written curriculum for the structured education programme, written presentation material for the educational sessions and participants' handouts, but also material for training for the educators who will deliver the programme.

The philosophy of the programme is based on patient empowerment. The structured group education programme will be based on psychological theories of learning including the Leventhal's common-sense theory, the dual-process theory, and the social learning theory. Similar to previous successful programmes in diabetes education and based on the experience gained by conducting the education programme "Living with type 2 diabetes" in our centre, the programme will be designed as a six-hour of education programme with a formal and informed curriculum. It will be offered in two three-hour sessions of teaching for 8-12 PCOS women at a time. Attendees will be encouraged to be accompanied by a person of their choice.

Initial thoughts on the curriculum and the format of the written material have been already discussed within our clinical and research team (Dr Papageorgiou, Professor Sathyapalan, Mrs Baldwin consultant endocrinologists, general practitioners and dietitian specialists/educators delivering the "Living with Diabetes" education programme for patients with type 2 diabetes) based on their experience and views expressed to them by women with PCOS. As such, the areas that will be covered in the structured education programme include:

* Thoughts and feelings of the participants around PCOS
* Understanding PCOS pathophysiology: what happens in the body
* Understanding the risk factors (e.g., obesity) and health risks associated with PCOS
* Emotional wellbeing and PCOS
* Management of PCOS symptoms -how to take control:

  * Pharmacological options (i.e., hormonal contraceptives, anti-androgens, and insulin sensitisers)
  * Lifestyle changes (i.e., basics of energy balance, healthy eating based on Eat well Plate, mindful eating, physical activity recommendations, practical advice).
* Planning for the future (e.g., family planning, screening for long-term conditions).

Importantly, the investigators are also going to conduct a patients' survey to find out what women with PCOS expect to gain from an educational programme addressing several aspects of PCOS. The investigators will use the collected data to further refine the aspects of PCOS that will be included in the final curriculum of the programme.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide signed informed consent before any study activity.
2. Women aged 18-50 years (inclusive), with a confirmed diagnosis of PCOS based on Rotterdam criteria.
3. Body mass index > 25 kg/m²

Exclusion Criteria:

1. Participants under 18 years or over 50 years old.
2. Participants who cannot adequately understand verbal and written explanations given in English.
3. Lack of mental capacity to give written consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female with PCOS aged between 18-50 years old will be involved
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
develop an evidence-based structured education programme for women with PCOS | 12 months
  Conducting a survey among women with PCOS to understand the service user's perspectives on the development of an educational programme for PCOS.
  The survey measures the need and knowledge about PCOS. The scales measures form 1 to 5. In which 1 is minimum or 5 is maximum. for example
  Information about PCOS
  1. Do you think you have enough knowledge about PCOS? Please circle the answer in the scale below
  1 2 3 4 5
Pilot the structured education programme | 12 months
  cognitive outcomes related to PCOS, monitor and evaluate the education process
  the post-pilot survey measures the satisfaction about the education session, the knowledge gained and the skills developed from the education session, the cognitive outcome and illness perception on a scale of 1 to 5 where 1 is minimum and 5 is maximum. for example
  How often do you think about your illness?
  1 2 3 4 5

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Academic diabetes, Endocrinology and metabolism, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make any identifiable participants data available to anyone. the final results will be published in one of the medical journals